CLINICAL TRIAL: NCT01443429
Title: A Pharmacokinetic Study of TRK-100STP -A Single Oral Administration Study in Japanese Patients With Renal Impairment as Compared to Subjects With Normal Renal Function
Brief Title: A Pharmacokinetic Study of TRK-100STP in Japanese Patients With Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Toray Industries, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 100CRS03
Record Dates: First submitted 2011-09-25; First posted 2011-09-29 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-03

CONDITIONS: Renal Impairment
Keywords: TRK-100STP; PK; beraprost sodium; Japanese males and females; Subjects with mild/moderate/severe patients; renal impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — beraprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- subjects with normal renal function (Experimental)
  Interventions: Drug: beraprost sodium(BPS)
- patients with mild renal impairment (Experimental)
  Interventions: Drug: beraprost sodium(BPS)
- patients with moderate renal impairment (Experimental)
  Interventions: Drug: beraprost sodium(BPS)
- patients with severe renal impairment (Experimental)
  Interventions: Drug: beraprost sodium(BPS)

INTERVENTIONS:
Drug: beraprost sodium(BPS)

SUMMARY:
The PK and safety profiles to be examined following a single oral administration of TRK-100STP (120 μg) under fasting conditions to patients with renal impairment and to subjects with normal renal function.

ELIGIBILITY:
Inclusion Criteria:

* The eGFR 1 day before study drug administration are stipulated as follows.
* Subjects with normal renal function : ≥90
* Patients with mild renal impairment : ≥60 to <90
* Patients with moderate renal impairment : ≥30 to <60
* Patients with severe renal impairment : ≥15 to <30

Exclusion Criteria:

* Patients on dialysis
* Patients who have a history of undergoing renal transplantation
* Patients with diabetes mellitus

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-08; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Composite of pharmacokinetic parameters of TRK-100STP such as maximum observed concentration (Cmax,pg/mL), area under the plasma concentration-time curve (AUC,pg·hr/mL), time at maximum concentration (Tmax,hr) and mean residence time (MRT,hr) | Up to 48hr

CONTACTS AND LOCATIONS:
Locations (1):
- Japan, Japan, Japan